CLINICAL TRIAL: NCT02187952
Title: Impact of Behavioral Feeding Intervention on Parent-Child Attachment in Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Amy K. Drayton, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-PAF07294
Record Dates: First submitted 2014-07-02; First posted 2014-07-11 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Pediatric Feeding Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Behavioral feeding intervention (Experimental): Behavioral feeding intervention will be conducted as usual. The intervention will not be altered for purposes of the study.
  Interventions: Behavioral: Behavioral feeding intervention
- Waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: Behavioral feeding intervention — Behavioral feeding intervention will include escape extinction.
  Arms: Behavioral feeding intervention

SUMMARY:
The primary objective of the proposed study is to determine whether behavioral feeding intervention impacts mother-child attachment in infants and toddlers with feeding problems. The investigators propose the following hypotheses:

* Behavioral feeding intervention will not significantly impact parent-child attachment.
* Behavioral feeding intervention will not significantly impact parent-child unstructured play interactions.
* Severity of feeding problems will decrease after behavioral feeding intervention is implemented.
* Behavioral feeding intervention will have either no significant effect or a significant positive effect on general child behavior.

ELIGIBILITY:
Inclusion Criteria:

Caregiver Based

* Mothers
* Conducts feeding intervention ≥75% of the time at home
* Understands and speaks English

Child Based

* 12-14 or 30-48 months old at initial assessment
* Clinically significant feeding problem
* Self-initiates movement
* Can be left alone in a room for 3 minutes
* Capable of initiating eye contact

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in attachment status | Enrollment, 6 months, 1 year
  The Strange Situation (SS) will be used to assess any changes in mother-child attachment status. The SS consists of a series of separations and reunions between a mother and her child.

SECONDARY OUTCOMES:
Change in infant social and emotional behavior | Enrollment, 6 months, 1 year
  Brief Infant Toddler Social Emotional Assessment (BITSEA) will be used to assess any changes in the social and emotional behavior of children who are 12-36 months of age.
Change in child externalizing and internalizing behavior. | Enrollment, 6 months, 1 year
  The Child Behavior Checklist will be used to assess any changes in the internalizing and externalizing behavior of children who are 1.5 to 5 years of age.
Change in maternal behavior when interacting with her child | Enrollment, 6 months, 1 year
  Mother-child dyads will be given toys and asked to play as they normally would for 10 minutes. The purpose of this measure is to detect any changes in parent-child interaction patterns that may be more sensitive to short-term intervention than attachment status.
Change in child feeding behavior. | Enrollment, 6 months, 1 year
  The Behavioral Pediatrics Feeding Assessment Scale (BPFAS) will be used to measure any changes in the feeding behavior of children.

CONTACTS AND LOCATIONS:
Overall Officials: Amy K Drayton, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States